CLINICAL TRIAL: NCT01712542
Title: Measurement of Intratumoral Concentration of the Nontoxic Natural Compound Curcumin in Glioblastoma Patients
Brief Title: Curcumin Bioavailability in Glioblastoma Patients
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Stephan Dützmann, M.D., Johann Wolfgang Goethe University Hospital
Other Study IDs: JohannWGUH_Curcumin-01
Record Dates: First submitted 2012-10-20; First posted 2012-10-23 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Patient Harboring Glioblastoma That Will Undergo Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tumor tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
Measuring the bioavailability of orally administered curcumin in the tumors of glioblastoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients harboring Glioblastoma
* Patient will undergo surgery

Exclusion Criteria:

* BMI > 30
* Liver and Kidney Function so compromised that medication is prescribed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients harboring Glioblastoma
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Concentration of Curcumin in Glioblastoma | At Tumor resection
  At the time of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Duetzmann, Principal Investigator — Goethe University
Locations (1):
- Department of Neurosurgery, Johann Wolfgang Goethe-University, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Senft C, Polacin M, Priester M, Seifert V, Kogel D, Weissenberger J. The nontoxic natural compound Curcumin exerts anti-proliferative, anti-migratory, and anti-invasive properties against malignant gliomas. BMC Cancer. 2010 Sep 14;10:491. doi: 10.1186/1471-2407-10-491. PMID 20840775